CLINICAL TRIAL: NCT04082897
Title: A Multi-Center, Open Label, Uncontrolled, Phase II Clinical Trial Evaluating the Safety and Efficacy of Venetoclax in Combination With Atezolizumab and Obinutuzumab in Richter Transformation of CLL
Brief Title: ObinutuzuMab AtezOlizumab and VenetocLax in RichTer transfOrmation
Acronym: MOLTO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOLTO
Record Dates: First submitted 2019-07-23; First posted 2019-09-10 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: CLL Transformation
Keywords: Richter Transformation; Safety; Efficacy; Obinutuzumab; Venetoclax; Atezolizumab
MeSH Terms: interventions — obinutuzumab; atezolizumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of Obinutuzumab, Atezolizumab and Venetoclax (Experimental): Obinutuzumab will be administered iv from cycle 1 to cycle 8 :
  * cycle1: 100 mg iv (day 1) and 900 mg iv (day 2) 1000mg iv (day 8 and day 15)
  * Cycle 2-8: 1000 mg iv on day 1
  Atezolizumab will be administered iv at 1.200 mg fixed dose from C1 to C18:
  * Cycles 1: day 2
  * Cycle 2-18: day 1
  Venetoclax will start from day 15 of cycle 1 on a weekly ramp-up basis:
  week 1: 20 mg (from day 15 cycle 1) week 2: 50 mg (from day 1 to day 7 cycle 2) week 3: 100 mg (from day 8 to day 14 cycle 2) week 4 200 mg (from day 15 to day 21 cycle 2) week 5: 400 mg (from day 1 cycle 3) venetoclax will be thereafter continued until day 21 of cycle 35
  Interventions: Drug: Obinutuzumab 25 MG/ML [Gazyva]; Drug: Atezolizumab 60 MG/ML [Tecentriq]; Drug: Venetoclax Oral Tablet

INTERVENTIONS:
Drug: Obinutuzumab 25 MG/ML [Gazyva] — Obinutuzumab will be administered from C1 to C8
Drug: Atezolizumab 60 MG/ML [Tecentriq] — Atezolizumab will be administered iv from C1 to C18
Drug: Venetoclax Oral Tablet — Venetoclax will be administered from day 15 cycle 1) until day 21 of cycle 35

SUMMARY:
This study is a multicenter, open-label, uncontrolled, phase II trial aimed to establish the safety and tolerability of venetoclax, atezolizumab and obinutuzumab combination in Richter Transformation of CLL.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, uncontrolled, phase II trial. Initial safety run phase is designed to establish the safety and tolerability of venetoclax, atezolizumab and obinutuzumab combination.

There is no dose-finding step. The doses of obinutuzumab and atezolizumab in lymphomas were previously clearly established in combination (Till BG et al. Blood 2015).

It has also been shown that in a balance between efficacy and toxicity, the recommended dose of venetoclax single-agent in Follicular Lymphoma (FL) and DLBCL was 800 mg daily (Davids MS et al. JCO 2017 ). The investigators chose the lower dose level (400 mg) for this study, also corresponding to the registered one for patients with CLL, in association with two other drugs. Nine patients having achieved 9 weeks (=3 cycles) of treatment (6 doses of obinutuzumab, 3 doses of atezolizumab, 7 weeks of venetoclax) or having discontinued treatment within the first 9 weeks of treatment will be enrolled in this cohort for safety profile. If one of these 9 patients prematurely discontinue at least one of study drugs for a reason other than safety (e.g. for disease progression), he/she will be replaced.

All AEs occurring during the course of the study will be captured, regardless of their intensity / grading. Grading of AEs will be completed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTC-AE), version 4.0. Based on known safety profile of the 3 drugs, some adverse events of special interest will be assessed. During the initial safety run phase, all haematological toxicities and immune-related toxicities whatever the grade, and grade ≥ 2 for other toxicities will be monitored and, in this case, safety review meeting will be organized with Independent Data Monitoring Committee (IDMC) members. In case of more than 3 non-infective and non-hematologic grade ≥4 adverse events in the initial safety run cohort that according to the experience of the investigators are considered related to the combination treatment, inclusions will be stopped and IDMC members will evaluate the possibility of an early enrollment termination.

The treatment schedule applied to the initial safety run cohort will be employed for the remaining patients.

The 9 patients from the safety run will be included in the efficacy analysis. A response evaluation according with Lugano criteria for aggressive lymphomas (Cheson et al. JCO 2014) will be performed at the end of the sixth cycle to define treatment efficacy and, in case of achievement of 16 responses, treatment will be considered successful.

The planned enrollment for this study is 28 patients.

Patients will receive 35 cycles of treatment:

* From cycle 1 to cycle 8 patients will receive a combination of obinutuzumab, atezolizumab and venetoclax
* From cycle 9 to cycle 18 patients will receive atezolizumab and venetoclax
* From cycle 19 to cycle 35 patients will receive venetoclax monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document
2. Signed Informed Consent
3. Confirmed diagnosis of chronic lymphocytic leukemia or small lymphocytic lymphoma as IW-CLL 2008 criteria (Hallek et al, 2008) with biopsy proven transformation to diffuse large B cell lymphoma (DLBCL), consistent with Richter's Syndrome
4. Age greater than or equal to 18 years
5. ECOG performance status <= 2
6. Patients must meet the following hematologic criteria at screening, unless they have significant bone marrow involvement of their malignancy confirmed on biopsy:

   * Absolute neutrophil count >=1000 cells/mm3 (1.0 x 10^9/L).
   * Platelet count >= 50,000 cells/mm3 (50 x 10^9/L) within 7 days of screening
   * Total hemoglobin > 9 g/dL (without transfusion support, unless anemia is due to marrow involvement of CLL)
7. Subject must have adequate coagulation, renal, and hepatic function, per laboratory reference range at screening as follows:

   * Activated partial thromboplastin time (aPTT) and International normalized ratio (INR) > 1.5 x ULN for patients not receiving therapeutic anticoagulation;
   * Creatinine <= 1.5 x ULN or creatinine clearance >= 50 mL/min based on Cockcroft-Gault formula;
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 2.5 × ULN;
   * Bilirubin <= 1.5 × ULN;
8. Subjects with Gilbert's Syndrome or resolving autoimmunohemolytic anemia may have a bilirubin up to 3.0 × ULN and are still eligible
9. Negative pregnancy tests as verified by the investigator prior to starting any treatment.

Exclusion Criteria:

1. Prior treatment for Richter transformation.
2. Prior treatment with obinutuzumab anti PD-1 or PDL-1 antibodies.
3. Prior treatment with venetoclax.
4. Hypersensitivity to obinutuzumab, venetoclax or atezolizumab or their formulation excipients.
5. Patients with the Hodgkin variant transformation of CLL.
6. Prolymphocytic transformation.
7. Patients with a previous history of indolent B cell malignancies other than CLL.
8. History of other malignancy other than CLL and Richter syndrome that could affect compliance with the protocol or interpretation of results with the exception of:

   1. Patients with curatively treated basal or squamous cell carcinoma or stage 1 melanoma of the skin or in situ carcinoma of the cervix
   2. Patients with a malignancy that has been treated with surgery alone with curative intent. Individuals in documented remission without treatment for > 2 years prior to enrollment may be included at the discretion of the Sponsor-Investigator.
   3. Low-risk prostate cancer on active surveillance.
9. Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results or that could increase risk to the patient, including renal disease that would preclude chemotherapy administration or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm).
10. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle1, Day1.
11. Clinically significant history of liver disease, including autoimmune hepatitis, current alcohol abuse, or cirrhosis.
12. Presence of positive PCR for hepatitis B, hepatitis C or positive hepatitis B surface antigen.
13. Patients with uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia.
14. History of active autoimmune disease.
15. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest CT scan at screening. History of radiation pneumonitis in the radiation field (fibrosis) is allowed.
16. Concurrent systemic immunosuppressant therapy within 28 days of the first dose of study drug.
17. Corticosteroids are allowed, but must be dosed at prednisone 30 mg (or equivalent) or lower prior to the start of chemotherapy.
18. Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
19. Known bleeding disorders (eg, von Willebrand's disease) or hemophilia.
20. Requires anticoagulation with vitamin K antagonists (e.g. phenprocoumon, warfarin)
21. History of human immunodeficiency virus (HIV) or active hepatitis C virus (HCV) or active hepatitis B virus (HBV).
22. Major surgery within 4 weeks of first dose of study drug.
23. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
24. Patients with infections requiring IV treatment (Grade 3 or 4) within the last 2 months prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the combination venetoclax, obinutuzumab and atezolizumab in terms of Overall Response Rate (ORR) | First 6 cycles of therapy (each cycle is 21 days)
  The treatment will be considered effective if the combination enables the achievement of a minimum of 67 % ORR at the end of the sixth cycle. Patients will be evaluated according to Lugano Criteria for aggressive lymphomas (Cheson et al. JCO, 2014). Residual underlying CLL may persist in node and/or marrow and still qualify as CR, denoting complete response of Richter Transformation (RT) to treatment (Hallek M et al. IwCLL Criteria Blood 2008).

SECONDARY OUTCOMES:
Safety (Incidence of Treatment-Emergent Adverse Events as assessed by NCI-CTCAE v4.0) of the combination venetoclax, obinutuzumab and atezolizumab | During the entire study duration (estimated to be 7 years)
  Incidence of Adverse Events (AE) and Serious Adverse Events (SAE) as measured per NCI-CTCAE v4.0;
Efficacy assessed by CRR of the combination venetoclax, obinutuzumab and atezolizumab | During the entire study duration (estimated to be 7 years)
  Assessment of the efficacy of the combination of obinutuzumab, atezolizumab and venetoclax with respect to Complete Remission Rate (CRR) defined as best response of CR
Efficacy assessed by DoR of the combination venetoclax, obinutuzumab and atezolizumab | During the entire study duration (estimated to be 7 years)
  Assessment of the efficacy of the combination of obinutuzumab, atezolizumab and venetoclax with respect to Duration of Response (DoR) defined as Time from first CR or PR to progressive disease (PD) or death
Efficacy assessed by PFS of the combination venetoclax, obinutuzumab and atezolizumab | During the entire study duration (estimated to be 7 years)
  Assessment of the efficacy of the combination of obinutuzumab, atezolizumab and venetoclax with respect to Progression Free Survival (PFS) defined as the time from enrolment to the first occurrence of disease progression or death, as determined by the investigator
Efficacy assessed by OS of the combination venetoclax, obinutuzumab and atezolizumab | During the entire study duration (estimated to be 7 years)
  Assessment of the efficacy of the combination of obinutuzumab, atezolizumab and venetoclax with respect to Overall Survival (OS) defined as the time from the enrolment to death from any cause.

CONTACTS AND LOCATIONS:
Locations (17):
- Italy (14):
  - Az. Ss.Antonio E Biagio E C.Arrigo - Osp.Civile Ss.Antonio E Biagio, Alessandria
  - Asst Papa Giovanni Xxiii, Bergamo
  - Azienda Ospedaliero-Universitaria Di Bologna, Bologna
  - Asst Degli Spedali Civili Di Brescia, Brescia
  - Asst Grande Ospedale Metropolitano Niguarda, Milan
  - Fond.Irccs "Istit.Naz.Le Tumori", Milan
  - Fondaz.Irccs Ca' Granda - Ospedale Maggiore Policlinico, Milan
  - Irccs S. Raffaele, Milan
  - Istituto Europeo Di Oncologia, Milan
  - Azienda Osped. Novara E Galliate - Osp. Maggiore Della Carita', Novara
  - Policlinico S. Matteo, Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Ao Citta' Della Salute E Della Scienza D- Osp.S. Giov.Battista Molinette, Torino
  - Asst Dei Sette Laghi, Varese
- Switzerland (3):
  - Istituto Oncologico della Svizzera Italiana (IOSI), Bellinzona
  - Luzerner Kantonsspital, Lucerne
  - Klinik für Hämatologie, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tedeschi A, Frustaci AM, Condoluci A, Coscia M, Chiarle R, Zinzani PL, Motta M, Gaidano G, Quaresmini G, Scarfo L, Catania G, Deodato M, Jones R, Tabanelli V, Griggio V, Stussi G, Calleri A, Pini K, Cairoli R, Zenz T, Signori A, Zucca E, Rossi D, Montillo M. Atezolizumab, venetoclax, and obinutuzumab combination in Richter transformation diffuse large B-cell lymphoma (MOLTO): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2024 Oct;25(10):1298-1309. doi: 10.1016/S1470-2045(24)00396-6. Epub 2024 Sep 10. PMID 39270702